CLINICAL TRIAL: NCT00133328
Title: A Morbi-Mortality and Remodeling Study With Valsartan in Patients With Hypertension and Cardiovascular Disease
Brief Title: A Morbidity-Mortality and Remodeling Study With Valsartan
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jikei University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHS2002
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2002-01

CONDITIONS: Hypertension; Ischemic Heart Disease; Congestive Heart Failure
Keywords: stroke; myocardial infarction; angina; renal damage
MeSH Terms: conditions — Hypertension; Myocardial Ischemia; Heart Failure; Stroke; Myocardial Infarction; Angina Pectoris | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
The JIKEI HEART Study has been designed to investigate whether concomitant treatment with valsartan, an angiotensin II receptor blocker (ARB), in addition to conventional treatment, will improve the prognosis of 3000 Japanese patients with cardiovascular diseases.

DETAILED DESCRIPTION:
Several recent clinical trials have demonstrated that angiotensin II receptor blockers (ARBs) have cardiovascular as well as renal protective effects. However, it is a problem that the number of Asian patients is very little in these trials. The researchers examine the treatment meaning by ARB about the prognosis of the patient who amalgamates either among high blood pressure, the ischemic heart disease, and congestive heart failures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension, ischemic heart disease and congestive heart failure

Exclusion Criteria:

* Pregnancy
* Severe renal damage
* Severe liver damage
* Acute myocardial infarction

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2002-01; Study Completion 2005-11

PRIMARY OUTCOMES:
stroke
new or recurrent transient ischemic attack
new or recurrent acute myocardial infarction
new occurrence or exacerbation of heart failure
new occurrence or exacerbation angina pectoris
dissecting aneurysm of the aorta
lower limb arterial obstruction
transition to dialysis
doubling of plasma creatinine (Cr) levels

SECONDARY OUTCOMES:
death from any cause
left ventricular hypertrophy
changes in ECG
proteinuria
B-type natriuretic peptide (BNP)
heart failure symptoms
heart failure syndrome (edema, rales on auscultation)
blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Seibu Mochizuki, MD., PhD, Study Chair — The Jikei University School of Medicine
Locations (1):
- The Jikei University School of Medicine, Tokyo, Japan

REFERENCES:
- [Result] Mochizuki S, Shimizu M, Taniguchi I, Kanae K, Yoshida S, Tajima N, Dahlof B; JIKEI HEART Study Group. JIKEI HEART Study--a morbi-mortality and remodeling study with valsartan in Japanese patients with hypertension and cardiovascular disease. Cardiovasc Drugs Ther. 2004 Jul;18(4):305-9. doi: 10.1023/B:CARD.0000041250.00079.84. PMID 15367828
- [Derived] Mochizuki S, Dahlof B, Shimizu M, Ikewaki K, Yoshikawa M, Taniguchi I, Ohta M, Yamada T, Ogawa K, Kanae K, Kawai M, Seki S, Okazaki F, Taniguchi M, Yoshida S, Tajima N; Jikei Heart Study group. Valsartan in a Japanese population with hypertension and other cardiovascular disease (Jikei Heart Study): a randomised, open-label, blinded endpoint morbidity-mortality study. Lancet. 2007 Apr 28;369(9571):1431-1439. doi: 10.1016/S0140-6736(07)60669-2. PMID 17467513 (Retraction: PMID 24012258 Lancet. 2013 Sep 7;382(9895):843)